CLINICAL TRIAL: NCT06133582
Title: Mood Awareness Psychotherapy Support - A Randomised Feasibility Trial of an Internet-Based Psychodynamic Treatment for University Students With Low Mood
Brief Title: Mood Awareness Psychotherapy Support
Acronym: MAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Linkoeping University (Other Government); Stockholm University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26049/001
Record Dates: First submitted 2023-11-08; First posted 2023-11-15 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Update January 2024: This trial has been transformed from a two arm randomised control trial to a single arm trial, due to challenges with recruitment. 51 participants have been successfully recruited and have now been invited to complete baseline measures. All participants will receive the intervention (the online therapy programme) once baseline data collection is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-Based Psychodynamic Psychotherapy (Experimental): Participants received the internet-based intervention for 10 weeks, supported by messages from their Therapeutic Support Worker.
  Interventions: Behavioral: Internet Based Psychodynamic Psychotherapy

INTERVENTIONS:
Behavioral: Internet Based Psychodynamic Psychotherapy — This is a 10-week intervention, delivered on a website called 'Iterapi' which was developed in Sweden. The programme involves creative and interactive web-based content- worksheets, audio, video, expressive writing exercises. Additionally, each participant is assigned a Therapeutic Support Worker (TSW). The TSW logs into the platform and views the questionnaires and other data provided by the participants that they are supporting. Each week, the TSW sends each of their participants a reflective message in response to the data they have provided when interacting with the programme over the last week. The participant can reply to this message.
  The principal objective of the iPDT intervention is to reduce depressive symptoms through the promotion of emotional awareness and emotional experience. The intervention is an affect-focused therapy and draws on Malan's Triangle of Conflict (Malan, 1995).

SUMMARY:
The aim of this single arm feasibility trial is to examine an internet delivered, self-help program for depression and anxiety, based on psychodynamic therapy. The study will evaluate the psychodynamic program with therapist support. The participants will be university students.

DETAILED DESCRIPTION:
Background: There appears to be an increase in mental health difficulties amongst higher education students in the UK. However, NHS services are over-stretched, and clients often experience long waits for treatment, during which time their symptoms may worsen. Internet-based therapies could be an important and accessible treatment option, particularly when provided within the context of the university, as this has the potential to provide timely treatment to those seeking help.

The majority of internet-based therapies use a Cognitive Behavioural Therapy framework. However, psychodynamic therapy has also been adapted to an internet-based format - often called 'iPDT'. One such iPDT programme was developed in Sweden for the treatment of adolescent depression. This is a self-guided programme, with therapist support. Clients 'chat' with their therapist once a week, for 30-minutes, using an instant-messaging platform on the therapy website. They can also send a-synchronous messages to their therapist, and the therapist can view the worksheets that client's complete on the therapy website.

This iPDT programme has been evaluated in two Randomised Controlled Trials, both of which showed it to be effective. Given the promising results of the Swedish iPDT programme, a research team at the Anna Freud Centre in the UK conducted a pilot study of an English-language version of the treatment; this pilot found evidence of a decrease in adolescents' symptoms of depression, and an improvement in emotion regulation, at the end of the 10-week treatment, with outcomes maintained at three month follow up.

At present, it is not known whether the iPDT programme would be accepted by, and effective for, participants without the weekly instant-messaging sessions. These 'chat sessions' are valued by many service users, but increase the cost and intensity of the programme. Furthermore, to date, the English-language version of the programme has not been tested with a university student population - young adults, rather than adolescents.

Study aims and design: This will be a single arm feasibility trial. The aim is to recruit approximately 50 university students with symptoms of depression and anxiety.

The aims of the study are to assess recruitment and retention rates of participants, including at three month follow up. To examine acceptability of the platform for the new target population, including levels of engagement with different elements of the treatment across the course of the intervention. The study will also explore indications of treatment efficacy. Additional exploratory analyses may be undertaken to explore moderators and mediators of change.

Participants will receive Internet Based Psychotherapy (iPDT). This is a 10-week intervention, delivered on the therapy website - called 'Iterapi' - which was developed at Linköping University in Sweden. The programme involves creative and interactive web-based content: worksheets, audio, video, expressive writing exercises. Additionally, each participant is assigned a Therapeutic Support Worker (TSW). The TSW logs into the platform and views the questionnaires and other data provided by the participants that they are supporting. Each week, the TSW sends each of their participants a reflective message in response to the data they have provided when interacting with the programme over the last week. The participant can reply to this message.

After completing the 10 week intervention, qualitative data will be collected via interviews with some participants to explore participants' experiences of the IPDT programme, in particular focussing on therapy process and their understandings of mechanisms of change, and of 'what works for whom'. Participants will also complete a set of follow up questionnaires 3 months after they complete the intervention.

The iPDT programme has 8 chapters. The principal objective of the iPDT intervention is to reduce depressive symptoms through the promotion of emotional awareness and emotional experience. The intervention is an affect-focused therapy and draws on Malan's Triangle of Conflict. Participants are invited to link their emotions to depressive symptoms, to challenge defences, regulate anxiety, and explore previously avoided feelings.

ELIGIBILITY:
Inclusion Criteria:

* score of 10 or more on the QIDS-SR

Exclusion Criteria:

* Under 18 years of age
* Not a current student at University College London (UCL)
* Previous diagnosis of: Bipolar disorder, any personality disorder, Psychosis / Schizophrenia, Post Traumatic Stress Disorder, intellectual disability
* Not being able to confidently read or write in English
* No access to a device which can access the internet
* Previous suicide attempts
* Current plans to attempt suicide
* Currently receiving psychological therapy
* Planning to begin psychological therapy during the duration of the intervention
* Starting new medication for mood, or using mood-medication inconsistently, over the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR) | Change from baseline to post-treatment (10 week) and follow up at 3 months after treatment (participants complete the measure weekly throughout the intervention)
  The 16-item QIDS-SR measures depressive symptoms. Scores range from 0-27, higher scores indicate more severe depression.

SECONDARY OUTCOMES:
Generalised Anxiety Disorder Questionnaire (GAD-7) | Change from baseline to post-treatment (10 week) and follow up at 3 months after treatment (participants complete the measure weekly throughout the intervention).
  The GAD-7 features seven items for assessing anxiety and screening for generalized anxiety disorder. Scores range from 0-21, higher scores indicate more severe anxiety.
Patient Health Questionnaire (PHQ-9) | Change from baseline to post-treatment (10 week) and follow up at 3 months after treatment. (Participants complete the measure at baseline, week 5, week 10, and follow up at 3 months).
  The PHQ-9 features nine items for assessing depression. Scores range from 0-27, higher scores indicate more severe depression.
Defences Questionnaire DMRS-SR-30 | Change from baseline to post-treatment (10 week) and follow up at 3 months after treatment. (Participants complete the measure at baseline, week 5, week 10, and follow up at 3 months).
  30-item self-rated measure of psychological defences

OTHER OUTCOMES:
The Working Alliance Inventory for guided Internet interventions (WAI-I) | Participants complete this measure at weeks 2, 3, 4, 5, 6, 7, 8, 9, & 10.
  12-item self-rated measure of working alliance. Scores range from 12-60, higher scores indicate a stronger alliance.
Depressive Experiences Questionnaire (DEQ English version) | Participants complete this at baseline, week 10, and 3 month follow up.
  66-item self-report questionnaire designed to differentiate between dependency and self-criticism in people experiencing depression.
Attitudes towards Psychological Online Interventions-the APOI | Participants complete this at baseline, week 10, and 3 month follow up.
  16-item self-report questionnaire designed to measure participants' attitudes towards and expectations of psychological online interventions. Higher scores indicate a more positive attitude towards psychological online interventions.
Relationship Styles Questionnaire | Baseline only.
  This is a self-report questionnaire designed to measure adult attachment style. Participants are presented with a short description of each attachment style (secure, fearful, preoccupied, dismissive). They first select which style best matches their own, and then rate each style on a likert scale from 1 - 7, where 1 is very unlike their relationship style, and 7 is very similar to their relationship style.
The Post Study System Usability Questionnaire (PSSUQ) - with minorly adapted wording to suit the therapy platform | Participants complete this in week 10
  16-item self-report questionnaire measuring participants' experience of using the therapy platform. Lower scores indicate greater satisfaction with the usability of the platform.
Interview | Participants complete this after week 10, before 3 month follow up.
  To explore participants' experiences of the IPDT programme, in particular focussing on therapy process and their understandings of mechanisms of change, and of 'what works for whom'.

CONTACTS AND LOCATIONS:
Overall Officials: Rose Mortimer, Study Chair — University College, London; Dominika Iluczyk, Study Chair — University College, London; Jakob Mechler, Study Chair — Stockholm University; Karin Lindqvist, Study Chair — Stockholm University
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindqvist K, Mechler J, Carlbring P, Lilliengren P, Falkenstrom F, Andersson G, Johansson R, Edbrooke-Childs J, Dahl HJ, Lindert Bergsten K, Midgley N, Sandell R, Thoren A, Topooco N, Ulberg R, Philips B. Affect-Focused Psychodynamic Internet-Based Therapy for Adolescent Depression: Randomized Controlled Trial. J Med Internet Res. 2020 Mar 30;22(3):e18047. doi: 10.2196/18047. PMID 32224489
- [Background] Mechler J, Lindqvist K, Carlbring P, Topooco N, Falkenstrom F, Lilliengren P, Andersson G, Johansson R, Midgley N, Edbrooke-Childs J, Dahl HJ, Sandell R, Thoren A, Ulberg R, Bergsten KL, Philips B. Therapist-guided internet-based psychodynamic therapy versus cognitive behavioural therapy for adolescent depression in Sweden: a randomised, clinical, non-inferiority trial. Lancet Digit Health. 2022 Aug;4(8):e594-e603. doi: 10.1016/S2589-7500(22)00095-4. Epub 2022 Jul 5. PMID 35803894
- [Background] Midgley N, Guerrero-Tates B, Mortimer R, Edbrooke-Childs J, Mechler J, Lindqvist K, Hajkowski S, Leibovich L, Martin P, Andersson G, Vlaescu G, Lilliengren P, Kitson A, Butler-Wheelhouse P, Philips B. The Depression: Online Therapy Study (D:OTS)-A Pilot Study of an Internet-Based Psychodynamic Treatment for Adolescents with Low Mood in the UK, in the Context of the COVID-19 Pandemic. Int J Environ Res Public Health. 2021 Dec 9;18(24):12993. doi: 10.3390/ijerph182412993. PMID 34948601
- [Derived] Mortimer R, Iluczyk D, Mechler J, Lindqvist K, Midgley N, Andersson G, Clements H. Experience of self-discovery and change in a psychodynamic internet delivered programme for university students experiencing low mood. Psychother Res. 2025 Aug 12:1-16. doi: 10.1080/10503307.2025.2538552. Online ahead of print. PMID 40791020